CLINICAL TRIAL: NCT01243801
Title: Phase 4 Study of Prevention of Persistent Postsurgical Pain After Thoracotomy Using Ketamine
Brief Title: Prevention of Persistent Postsurgical Pain After Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Beatriz Tena, Dr Tena, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BTB-10
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Persistent Pain; Postoperative Hyperalgesia
Keywords: chronic pain; persistent postsurgical pain; hyperalgesia; ketamine; quantitative sensory testing
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative; Hyperalgesia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epidural ketamine (Active Comparator): * Bolus of epidural ketamine during the induction of anesthesia
  * Epidural infusion of ketamine during the first 48 h after surgery
  Postoperative analgesia: Epidural "Patient Controlled Analgesia" with ropivacaine and fentanyl
  Interventions: Drug: Ketamine
- Intravenous ketamine (Active Comparator): * Bolus of intravenous ketamine administered during the induction of anesthesia
  * Intravenous infusion during the first 48 hours after surgery
  Postoperative analgesia: Epidural "Patient Controlled Analgesia" with ropivacaine plus fentanyl
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Postoperative analgesia: Epidural "Patient Controlled Analgesia" with ropivacaine and fentanyl
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Intravenous ketamine 0.5mg/kg(induction of anesthesia)and 0.25 mg/kg/h for 48h Epidural Ketamine 0.5 mg/kg(induction of anesthesia)and 0.25 mg/kg/h for 48h

SUMMARY:
Postthoracotomy acute pain is followed by persistent postsurgical pain in 20-30% of the patients, defined as pain that lasts more than 3-6 months after surgery. Acute pain and hyperalgesia around the surgical wound are some of the risk factors associated to the development of chronic pain. Ketamine, as a NMDA antagonist mainly at spinal level, might reduce periincisional hyperalgesia and persistent postsurgical pain after thoracotomy. Therefore, the investigators hypothesized that continuous ketamine infusion at subanesthetic dose would potentiate epidural ropivacaine and fentanyl-induced analgesia after thoracotomy, reduce periincisional hyperalgesia and long-term postoperative pain. To test these hypothesis, the investigators administered a low dose of intravenous ketamine or epidural ketamine or placebo to patients who received an epidural infusion of ropivacaine and fentanyl for postthoracotomy pain.

DETAILED DESCRIPTION:
Chronic pain is a frequent complication after common surgical procedures such as amputation, mastectomy or thoracotomy. A rate between 20 and 60% of patients undergoing thoracotomy are reported to develop long-lasting pain.

The causes of chronic pain after surgery are not fully known but several risk factors have been identified including pre and postoperative pain, nerve injury during surgery and physicological and genetic factors. The observed symptoms of allodynia and hyperalgesia in the periincisional area and evidence of intercostal nerve injury due to rib retraction during surgery suggest a neuropathic aetiology.

Excitatory neurotransmitters, acting through N-metil-aspartate receptor, have been recently postulated to play an important role in the development and maintenance of pathologic pain states. In experimental pain research, NMDA receptor antagonists reduced wind-up and central sensitization. Ketamine is one of the few NMDA antagonists available in clinical practice that, administered at subanesthetic doses, would inhibit the spinal processing of nociceptive input.

It has been proposed that analgesic drugs might more adequately prevent central sensitization when administered during the entire period of high-intensity noxious stimulation.

Therefore, the investigators hypothesized that continuous ketamine infusion would potentiate epidural ropivacaine and fentanyl-induced analgesia after posterolateral thoracotomy or minithoracotomy, reduce periincisional hyperalgesia and long-term postoperative pain. To test these hypothesis, the investigators administered a low dose of intravenous or epidural ketamine or placebo to patients who received an epidural infusion of ropivacaine and fentanyl for postthoracotomy pain.

The Institutional Review Board of the hospital approved this study, and each patient gave written informed consent. The investigators planned to enroll 90 patients who were scheduled to undergo posterolateral thoracotomy or minithoracotomy in this double-blind, controlled, randomized study. Patients who met the inclusion and exclusion criteria would be included and assigned to one of the three groups by a computer-generated schedule. Patients, nurses in charge of postoperative care, and staff members, who inform the patient performed analgesia, and collected data are blinded to the group.

The day before surgery patients are instructed on the use of Patient Controlled Analgesia pump, Visual Analogue Scale (VAS) and the Quantitative Sensory Testing. Subjective tests (VAS, neuropathic pain symptom inventory, pain catastrophizing scale) and QST are also performed the day before surgery.

Anesthetic management is standardized to all study patients. Premedication with sublingual diazepam (5-10 mg) is administered 2 hours before surgery. A thoracic epidural catheter is placed before induction through the T7-8 interspace. General anesthesia is induced by fentanyl (3 mcg/kg), propofol (2mg/kg) and cisatracurium (0.15 mg/kg). A double-lumen endobronchial tube is placed to perform differential one-lung ventilation. The left radial arteria is secured for arterial pressure monitoring and arterial blood sampling. Monitoring included electrocardiography, haemoglobin oxygen saturation, end-tidal carbon dioxide tension and invasive arterial pressure. A bolus of ketamine or placebo, intravenous or epidurally, according to the group of study is administered before skin incision. The study drug is prepared and placed by a nurse who does not participate in the anesthesia or evaluation of postoperative pain. Anesthesia is maintained by sevoflurane 1.5-2%, fentanyl and cisatracurium titrated according to the patients´needs. At the end of the skin closure, 5-7 ml of ropivacaine 0.2% is administered epidurally followed by epidural infusion of ropivacaine 0.15% and fentanyl 2mcg/ml and epidural or intravenous infusion of ketamine or placebo according to the group. Patients are extubated in the operating room and transferred to the postanesthesia care unit.

Epidural infusion is maintained for 48 hours at a rate of 3-6ml/h, boluses of 2-3 ml are allowed every 20 minutes.The protocol for rescue analgesia consisted of the first administration of iv metamizol 2g per 8 hours. The second rescue analgesia line consisted of the adjunction of subcutaneous methadone 3-6 mg per 8 hours. Patients remained in the postanesthesia care unit for 24 hours. Pain at rest and on coughing is assessed with VAS at 1-4-8-12-24-72 hours. Side effects including cognitive effects such as nightmares or hallucinations, blurred vision, sedation (not arousable except by persisting verbal or tactile stimulation), or haemodynamic effects (hypertension over 20% their basal values). Subjective test and QST are performed at 72h, 7 day, 3 and 6 months after surgery.

The investigators considered 30 patients per group in order to obtain 3 points of difference of the ratio between the hyperalgesia area and the incision length, considering a SD of differences of 3.5, type I error of 0.05 and statistical power of 0.9.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old submitted to thoracotomy or minithoracotomy expected to be extubated in the operating room

Exclusion Criteria:

* Allergy or intolerance to ketamine, local anesthetics or opioids
* Chronic preoperative pain
* Chronic opioid treatment
* Drug addiction
* Polyneuropathy
* Ischemic cardiopathy
* Psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-09; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from subjective pain scales: Visual Analogical Scale, Neuropathic Pain Symptoms Inventory, Catastrophism Scale | -1day, 3 days, 7 days, 3 months, 6 months
  Pain measured with these subjective scales are assessed preoperatively (-1 day) and 3, 7 days, 3 and 6 months after surgery
Change from hyperalgesia periincisional area | -1day, 3day,7day,3 months, 6 months
  Hyperalgesia is measured with von Frey monofilaments, electronic von frey and electric brush around the surgical incision and in a separate area (thigh)

SECONDARY OUTCOMES:
Adverse effects | any time until 6 months
  Any adverse effects related to the use of ketamine (cognitive effects, visual effects, haemodynamic effects or sedation effects)

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Tena, MD, Principal Investigator — Hospital Clinic of Barcelona; Carmen Gomar, PhD, Study Director — Hospital Clinic of Barcelona; Irene Rovira, PhD, Study Chair — Hospital Clinic of Barcelona; Maria J Jimenez, PhD, Study Chair — Hospital Clinic of Barcelona; Guillermina Fita, PhD, Study Chair — Hospital Clinic of Barcelona; Samuel Garcia, MD, Study Chair — Hospital Clinic of Barcelona; Jordi Perez, PhD, Study Chair — Hospital Clinic of Barcelona; Daniel Poggio, MD, Study Chair — Hospital Clinic of Barcelona; Jose Rios, Study Chair — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Department Anesthesia. Hospital Clinic Barcelona, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona

REFERENCES:
- [Background] De Kock MF, Lavand'homme PM. The clinical role of NMDA receptor antagonists for the treatment of postoperative pain. Best Pract Res Clin Anaesthesiol. 2007 Mar;21(1):85-98. doi: 10.1016/j.bpa.2006.12.006. PMID 17489221
- [Background] Suzuki M, Haraguti S, Sugimoto K, Kikutani T, Shimada Y, Sakamoto A. Low-dose intravenous ketamine potentiates epidural analgesia after thoracotomy. Anesthesiology. 2006 Jul;105(1):111-9. doi: 10.1097/00000542-200607000-00020. PMID 16810002